CLINICAL TRIAL: NCT06640907
Title: Universal Prevention of Maternal Perinatal Mental Disorders and Its Implementation as Normalized Routine Practice (e-Perinatal): Pilot Randomized Control Trial (WP2)
Brief Title: Feasibility Study and Pilot Hybrid Effectiveness-Implementation Trial for the Universal Prevention of Maternal Perinatal Mental Disorders as Normalized Routine Practice (e-Perinatal Pilot)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Seville (Other)
Collaborators: Health Service of Andalucia (Other Government); Junta de Andalucia (Other Government)
Responsible Party: Principal Investigator, Emma Motrico, Research Fellow in Psychology, University of Seville
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SICEIA-2024-001659; 101042139 (Other Grant/Funding Number: European Research Council (ERC))
Record Dates: First submitted 2024-10-08; First posted 2024-10-15 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Perinatal Depression; Perinatal Anxiety
Keywords: Depression; Anxiety; Perinatal; Well-being; Prevention; mHealth
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Cluster-randomized hybrid type 1 controlled trial
Who Masked: Outcomes Assessor
Masking Description: Data analysts will also be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental)
  Interventions: Behavioral: e-Perinatal personalized mHealth intervention integrated into routine maternal care
- Control group (Active Comparator)
  Interventions: Other: Standard routine maternal care with general perinatal health information

INTERVENTIONS:
Behavioral: e-Perinatal personalized mHealth intervention integrated into routine maternal care — The e-Perinatal intervention combines a personalized mobile health (mHealth) app with targeted training for healthcare professionals to support perinatal mental health within routine maternal care. Participants allocated to the intervention arm will use the app for a period of two months. The app offers psychoeducational content, video-guided physical activities, mindfulness exercises, mood-tracking tools, personalized recommendations through a rule-based algorithm, and social-community features. Healthcare professionals assigned to the intervention arm receive specialized training to integrate the app into their daily practice, enhancing their ability to promote and support mental health during the perinatal period.
  Arms: Intervention group
Other: Standard routine maternal care with general perinatal health information — Standard maternal care as routinely provided by the Andalusian public healthcare system (Spain). This includes scheduled visits with midwives, nurses, and pediatrician for maternal and infant health monitoring, as well as access to childbirth education programmes. Participants also receive monthly psychoeducational emails (two months) containing general information on perinatal mental health, pregnancy, and infant development. Healthcare professionals in this arm do not receive specialized training in perinatal mental health or in the use of digital interventions, and participants do not have access to the e-Perinatal app.
  Arms: Control group

SUMMARY:
This study is part of the e-Perinatal project, funded by the European Research Council. This research project will follow the first three phases recommended by the Medical Research Council (MRC) framework for the development and evaluation of complex interventions (Skivington et al., 2021).

The primary aim is to evaluate the feasibility and acceptability of implementing an innovative, personalized mobile health (mHealth) intervention designed for the universal prevention of perinatal mental disorders. Using a pilot, two-arm, cluster-randomized hybrid type 1 clinical trial, the study will assess key implementation outcomes and preliminary effectiveness indicators. The findings will inform the design of a future large clinical trial, intending to evaluate the effectiveness, cost-effectiveness, and implementation of the intervention as part of maternal care.

DETAILED DESCRIPTION:
This pilot clinical study investigates the feasibility, acceptability, and preliminary implementation and effectiveness of the e-Perinatal app, an innovative, personalized mobile health (mHealth) intervention designed for the universal prevention of perinatal mental disorders. The study will be conducted as a two-arm, cluster-randomized, hybrid type 1 trial within routine maternal care settings in primary healthcare centers in Andalusia, Spain. Participants will include pregnant and postpartum women (up to five months postpartum) and their partners. Primary healthcare centers will be randomized to either the intervention or control arm.

The primary objective is to evaluate the feasibility of integrating the e-Perinatal app into routine maternal care. Secondary objectives include assessing the acceptability of the intervention among women, partners, and healthcare professionals and exploring preliminary effectiveness outcomes, such as the incidence of perinatal depression and anxiety in women, changes in depressive and anxiety symptoms in both women and their partners, and potential impacts on infant health and development.

The study hypothesizes that the e-Perinatal intervention will be feasible and acceptable for pregnant and postpartum women, their partners, and healthcare professionals involved in routine maternal care.

Participants will be recruited from primary healthcare centres and allocated by cluster randomization to either the intervention group, which will receive the e-Perinatal app along with standard maternal care, or the control group, which will receive standard maternal care and monthly psychoeducational emails.

ELIGIBILITY:
Inclusion criteria for mothers:

* Must receive an invitation to participate from a healthcare professional at one of the participating primary healthcare centers
* Must be pregnant for at least 16 weeks or have given birth within the last 5 months at the time of enrollment
* Must be at least 18 years old
* Must have access to a mobile phone and internet connection
* Must be able to read, write, and understand Spanish
* Must have a personal email account

Inclusion criteria for partners (or significant others):

* Must receive an invitation to participate from a woman already enrolled in the study
* Must be at least 18 years old
* Must have access to a mobile phone and internet connection
* Must be able to read, write, and understand Spanish
* Must have a personal email account

Exclusion criteria for mothers:

* Meet diagnostic criteria for anxiety or depression, as determined by a structured clinical interview
* Be on a waiting list or currently receiving psychological or pharmacological treatment for any mental health or substance use condition

Exclusion criteria for partners (or significant others):

* There are no exclusion criteria for partners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2025-05-02 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the intervention | Measured at baseline and postintervention (2 months after baseline)
  Calculation of participation rate, recruitment rate, and retention rate (follow-up rate) at all assessment points. Assessment method: Registration and follow-up records.
Early acceptability | Measured at enrollment
  Number of eligible women and partners who agree to participate. Assessment method: Consent forms.
Final acceptability | Measured at postintervention (2 months after baseline)
  Evaluation of how appropriate, satisfactory, and feasible the intervention is after its implementation. Assessment method: Surveys and semi-structured interviews based on the Normalization Process Theory.

SECONDARY OUTCOMES:
Adoption | Measured before recruitment
  Proportion of Primary Health Care (PHC) professionals who express their willingness to participate in the study among the total of potential professionals prior to the start of the intervention. Assessment method: Registration records.
Fidelity | Measured at postintervention (2 months after baseline)
  Measures adherence to the study protocol by PHC professionals. Assessment method: Surveys.
Early appropriateness | Measured at enrollment
  Number of eligible women and number of partners invited to participate by women. Assessment method: Consent forms and recruitment records.
Final appropriateness | Measured at postintervention (2 months after baseline)
  Suitability and relevance of the intervention for the target population and context. Assessment method: Semi-structured interviews based on the Normalization Process Theory.
Cumulative incidence of maternal perinatal depression and maternal perinatal anxiety | Measured at enrollment and postintervention (2 months after baseline)
  Measurement of the incidence of maternal perinatal depression and anxiety. Assessment method: The Mini International Neuropsychiatric Interview (MINI).
Depressive symptoms | Measured at enrollment, postintervention (2 months after baseline), and follow-up (1 month after postintervention)
  Changes in depressive symptoms. Assessment method: The Edinburgh Postnatal Depression Scale (EPDS), a 10-item self-report measure. Each item is scored from 0 to 3, with higher scores indicating more severe depressive symptoms.
Anxiety symptoms | Measured at enrollment, postintervention (2 months after baseline), and follow-up (1 month after postintervention)
  Changes in anxiety symptoms. Assessment method: The General Anxiety Questionnaire (GAD-7), a 7-item self-report measure. Each item is scored from 0 to 3, with higher scores indicating more severe anxiety symptoms.
Postnatal post-traumatic stress | Measured at baseline
  Presence of post-traumatic stress symptoms and clinical disorder in women or their partners after childbirth. Assessment method: Assessed using City Birth Trauma Scale (City-BiTS), a 31-item self-report measure. Some items are scored from 0 to 3 and others from 0 to 2, with higher scores indicating greater severity of postnatal post-traumatic stress.
Well-being | Measured at baseline, postintervention (2 months after baseline), and follow-up (1 month after postintervention)
  Changes in subjective well-being. Assessment method: The Well-Being Index (WHO-5), a 5-item self-report measure. Each item is scored from 0 to 5, with higher scores indicating better subjective well-being.

OTHER OUTCOMES:
Organizational readiness for implementing change | Measured before recruitment
  Organization's readiness for implementing changes in usual care. Assessment method: The Organizational Readiness Implementing Change (ORIC), a 12-item self-report measure. Each item is scored from 1 to 5, with higher scores indicating greater readiness for implementing change.
App quality | Measured at postintervention (2 months after baseline)
  Objective and subjective quality, and the perceived impact of the application. Assessment method: The User Version of the Mobile Application Rating Scale (u-MARS), a 26-item self-report measure. Each item is scored from 1 to 5, with higher scores indicating better app quality.
Implementation process | Measured at postintervention (2 months after baseline)
  App implementation process from the perspective of healthcare professionals involved in implementing complex interventions. Assessment method: The Normalization Measure Development Questionnaire (NoMAD), a 20-item self-report measure. Each item is scored from 1 to 5, with higher scores indicating more effective implementation processes.
Barriers and facilitators | Measured at postintervention (2 months after baseline)
  Identifies barriers and facilitators impacting the integration of the intervention into routine healthcare, drawing from the experiences of users and healthcare professionals. Assessment method: Semi-structured interviews following the Normalization Process Theory (NPT) framework
PHC characteristics | Measured before recruitment
  Size of the population where the PHC is located and number of PHC professionals. Assessment method: Questionnaire developed by the research team
Reasons for dropout | Measured at postintervention (2 months after baseline)
  Number and reasons (e.g., experienced miscarriage or stillbirth, lack of engagement with the app) for dropout among women and their partners. Assessment method: Records and semi structured interviews.
Antenatal and postnatal risks | Measured at baseline
  Measures both antenatal and postnatal risk factors. Assessment method: The Antenatal Risk Questionnaire (ANRQ-R), a 11-item self-report measure. Some items are scored from 1 to 5 and others are scored on categorical scale, with higher scores indicating greater risk.
Maternal antenatal attachment | Measured at baseline
  Measures the level of maternal antenatal attachment to the baby. Assessment method: The Maternal Antenatal Attachment Scale (MAAS), a 19-item self-report measure. Each item is scored from 1 to 5, with higher scores indicating stronger maternal antenatal attachment.
Paternal antenatal attachment | Measured at baseline
  Measures the level of paternal antenatal attachment to the baby. Assessment method: The Paternal Antenatal Attachment Scale (PAAS), a 16-item self-report measure. Each item is scored from 1 to 5, with higher scores indicating stronger paternal antenatal attachment.
Maternal postnatal attachment | Measured at baseline
  Measures the level of maternal postnatal attachment to the baby. Assessment method: The Maternal Postnatal Attachment Scale (MPAS), a 19-item self-report measure. Each item is scored from 1 to 5, with higher scores indicating stronger maternal postnatal attachment.
Paternal postnatal attachment | Measured at baseline
  Measures the level of postnatal attachment to the baby in both mothers and fathers. Assessment method: The Paternal Postnatal Attachment Scale (PPAS), a 19-item self-report measure. Each item is scored from 1 to 5, with higher scores indicating stronger paternal postnatal attachment.
Infant temperament | Measured at baseline
  Measures various aspect of infant temperament. Assessment method: The Infant Behavior Questionnaire-Revised Short Form (IBQ-R SF), a 37-item self-report measure. Each item is scored from 1 to 7, with higher scores indicating a higher frequency of the specified temperament behavior.
Coparenting dynamics | Measured at baseline
  Measures the dynamics of coparenting relationships. Assessment method: The Coparenting Relationship Scale (CRS), a 14-item self-report measure. Each item is scored from 0 to 6, with higher scores indicating more positive coparenting dynamics.
Parental role perception | Measured at baseline
  Measures parents' perception of their competence in the parental role. Assessment method: The Parental Sense of Competence scale (PSOC), a 21-item self-report measure. Each item is scored from 1 to 6, with higher scores indicating a stronger sense of parental competence.
Infant development | Measured at baseline
  Measures various developmental milestones in infants.
Partnership quality | Measured at baseline
  Measures the quality of the marital or partnership relationship. Assessment method: The Quality of Marriage Index (QMI), a 6-item self-report measure. Some items are scored from 1 to 7 and others from 1 to 10, with higher scores indicating better relationship quality.
Sleep quality | Measured at baseline
  Measures the quality of sleep among participants. Assessment method: The Pittsburgh Sleep Quality Index (PSQI), a 19-item self-report measure. Some items are scored from 0 to 3 and some on a categorical scale, with higher scores indicating poorer sleep quality.
Life quality | Measured at baseline
  Measures the overall quality of life. Assessment method: The European Quality of Life-5 Dimensions-5 Levels (EuroQol-5D-5L), a 5-item self-report measure. Each item is scored from 1 to 5, with higher scores indicating worse quality of life.
Maternal physical activity levels | Measured at baseline
  Measures physical activity levels in pregnant women and mothers. Assessment method: The Pregnancy Physical Activity Questionnaire (PPAQ), a 33-item self-report measure. Each item is scored from 0 to 5, with higher scores indicating higher levels of physical activity.
Paternal physical activity levels | Measured at baseline
  Measures physical activity levels in fathers. Assessment method: The International Physical Activity Questionnaire (IPAQ), a 7-item self-report measure. Each item is scored on a categorical scale, with higher scores indicating higher levels of physical activity.
Physical condition | Measured at baseline
  Measures overall physical condition and the main components (i.e., cardiorespiratory fitness, muscular strength, speed-agility, and flexibility) in pregnant women and mothers. Assessment method: The International FItness Scale (IFIS), a 5-item self-report measure. Each item is scored from 1 to 5, with higher scores indicating better physical condition.
Mood state | Measured at baseline
  Measures positive and negative affect states. Assessment method: The Positive and Negative Affect Schedule (PANAS), a 20-item self-report measure. Each item is scored from 1 to 7, with higher scores indicating a higher frequency of the specified temperament behavior.
Basic psychological needs | Measured at baseline
  Measures the satisfaction and frustration of basic psychological needs. Assessment method: The Basic Psychological Need Satisfaction and Frustration Scale - Short Form (BPNSFS), a 12-item self-report measure. Each item is scored from 1 to 5, with higher scores indicating a higher need satisfaction (i.e., need satisfaction subscale) or a higher need frustration (i.e., need frustration subscale).
Economic data | Measured at postintervention (2 months after baseline)
  Measures healthcare service utilization and sick leave days over the previous year among participating women.
  Assessment method: a post hoc semi-structured interview that collects information on emergency visits, hospital admissions, primary care visits (e.g., nurse, midwife, social worker), secondary care visits, and consultations with specialists.

CONTACTS AND LOCATIONS:
Locations (1):
- Primary Health Care Center Mairena del Aljarafe - Ciudad Expo, Mairena del Aljarafe, Seville, Spain

IPD SHARING:
Plan to Share IPD: No